CLINICAL TRIAL: NCT06583603
Title: Identifying Barriers to Implementing Sensory Strategies in the Classroom Setting: a Teacher's Perspective
Brief Title: Identifying Barriers to Implementing Sensory Strategies in the Classroom Setting
Status: Not yet recruiting | Type: Observational
Sponsor: Bay Path University (Other)
Responsible Party: Principal Investigator, Allison Niemiec, Occupational Therapist, Bay Path University
Other Study IDs: BPU
Record Dates: First submitted 2024-07-31; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Sensory Disorder
Keywords: sensory processing; classroom setting; sensory strategies or sensory treatment; maladaptive behaviors or challenging behaviors
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Survey: 17-item electronic survey will be administered via google docs
  Interventions: Behavioral: Barriers to Implementing Sensory Strategies Survey

INTERVENTIONS:
Behavioral: Barriers to Implementing Sensory Strategies Survey — Survey, see arm description

SUMMARY:
The goal of this clinical trial is to determine barriers to implementing sensory strategies in the classroom setting as well as potential supports needed in teachers and paraprofessionals 18 years and older who are actively working in the classroom setting. The main questions it aims to answer are:

1. What are common themes that limit classroom staff from implementing sensory strategies within the classroom setting?
2. What support do classroom staff need from an occupational therapist to feel confident in implementing sensory strategies within their classroom?

Participants will be asked to participate in a 17-item electronic survey via Google Forms. They will be asked to provide informed consent prior to participating.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Active teacher or paraprofessional working in the classroom

Exclusion Criteria:

* Younger than 18 years old
* Teachers or paraprofessionals no longer actively working in the classroom setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Teachers and paraprofessionals who are 18 years and older and are actively working in the classroom setting
Sampling Method: Non-Probability Sample
Enrollment: 365 (Estimated)
Dates: Start 2024-09-06 (Estimated); Primary Completion 2024-10-06 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Barriers to implementing sensory strategies in the classroom setting | 13 weeks
  Survey will be dispersed via email and Facebook groups. Survey will be on google docs.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Niemiec, Principal Investigator — Bay Path University

IPD SHARING:
Plan to Share IPD: No